CLINICAL TRIAL: NCT06219551
Title: The Effect of Supporting Routine Smoking Cessation Interventions With Whatsapp-mediated Motivational Information on Smoking Cessation Success in Active Smokers With Inflammatory Rheumatic Diseases: A Randomized Controlled Study
Brief Title: Smoking Cessation Support for Patients With Rheumatologic Diseases Via WhatsApp
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enough participants included to the study.
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dilek KARADOĞAN, Associated Professor, M.D, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRW
Record Dates: First submitted 2023-12-13; First posted 2024-01-23 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Tobacco Use Cessation
Keywords: tobacco cessation; rheumatologic diseases; smoking cessation support
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: Randomized controlled, paralel arm, prospective cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (Active Comparator): Usual care arm, smoker patients with rheumatologist diseases will be implemented brief smoking cessation interventions and referred to quit lines or smoking cessation services and also directly contacted to get an appointment from the cessation clinic.
  Interventions: Other: Mobile messages via What's App
- Intervention (Experimental): The intervention arm, smoker patients with rheumatologist diseases will be implemented brief tobacco cessation interventions and directly contacted to get an appointment from cessation clinic and will be send periodically motivational and informative text messages regarding tobacco cessation via WhatsApp.
  Interventions: Other: Mobile messages via What's App

INTERVENTIONS:
Other: Mobile messages via What's App — The information article that was prepared by taking the opinions of academics experienced in adult education, and were prepared as a video by the primary Rheumatologist who performs the randomization and will be shared in the Whatsapp group as information. Additionally, information will be provided once a week regarding the appointment date of the smoking cessation clinic.

SUMMARY:
Smoking cessation support for patients with rheumatologist diseases is an underestimated issue. In the previous prospective cohort study the investigators determined that with the brief cessation interventions 63.5% of smokers with rheumatologic diseases were willing to quit and the rest 36.4% were not willing. Among the willing group the highest quit rate was detected in the group that admitted to smoking cessation clinic. Therefore to increase the willingness to quit as well as to increase the Access to evidence based tobacco cessation support using new comminication technologies can be relevant. Investigators' aim in this study is to examine the effect of including WhatsApp in the routine smoking cessation practices on the quitting success of active smokers with rheumatic diseases who apply to the Rheumatology outpatient clinic.

DETAILED DESCRIPTION:
In this randomized controlled study, the sample will be randomly divided to 2 arms. In one arm, usual care arm, smoker patients with rheumatologist diseases will be implemented brief smoking cessation interventions and referred to quit lines or smoking cessation services and also directly contacted to get an appointment from the cessation clinic. In the other arm, the intervention arm, smoker patients with rheumatologist diseases will be implemented brief tobacco cessation interventions and directly contacted to get an appointment from cessation clinic and will be send periodically motivational and informative text messages regarding tobacco cessation via WhatsApp.

Primary outcome measures will be the quit rate of both arms at 3rd, 6th and 12th month.

Secondary outcomes will be access to evidence based smoking cessation support, admission rate of smoking cessation clinic and treatment use duration of cessation medications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients applying to the rheumatology outpatient clinic
2. Those aged 18 and over
3. Those who are active smokers
4. Those diagnosed with inflammatory rheumatic disease
5. Those who gave informed written consent to participate in the study

Exclusion Criteria:

1. Those with active psychiatric disease diagnoses such as psychosis, major depression, schizophrenia among their current diagnoses
2. Those with cognitive dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of participants with successful quit attempt | 3-6 and 12 months after the randomization
  Successful quitter: sustained abstinence since the target quit date will be asked and validated by exhaled breath carbon monoxide measure.

SECONDARY OUTCOMES:
Access to evidence based cessation support | Within one year after the randomization
  Admitters to cessation clinics

CONTACTS AND LOCATIONS:
Overall Officials: Osman Cüre, M.D, Principal Investigator — Recep Tayyip Erdoğan University Department of Rheumatology
Locations (1):
- Recep Tayyip Erdoğan University, Training and Research Hospital, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheung YT, Chan CH, Lai CK, Chan WF, Wang MP, Li HC, Chan SS, Lam TH. Using WhatsApp and Facebook Online Social Groups for Smoking Relapse Prevention for Recent Quitters: A Pilot Pragmatic Cluster Randomized Controlled Trial. J Med Internet Res. 2015 Oct 22;17(10):e238. doi: 10.2196/jmir.4829. PMID 26494159
- See also: An example of a comprehensive approach to increase the access to evidence-based tobacco cessation support for smokers with rheumatic diseases — http://www.populationmedicine.eu/pdf-175000-97034?filename=An%20example%20of.pdf